CLINICAL TRIAL: NCT05294263
Title: Varenicline for Comorbid Tobacco and Cannabis Use in Veterans
Brief Title: Varenicline for the Treatment of Cannabis and Tobacco Use Disorders in Veterans
Acronym: Vet Cat
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Despite the numerous approaches below, we have not been successful in identifying a recruitment pathway that would ensure feasibility of study continuation. We have had multiple meetings with CSR&D leadership to discuss our study progress
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NURA-004-21S; I01CX002357 (NIH)
Record Dates: First submitted 2022-02-09; First posted 2022-03-24 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Tobacco Use Disorder; Cannabis Use Disorder
Keywords: Nicotine; Smoking; Tobacco Use Disorder; Cannabis; Marijuana Abuse; Marijuana Smoking; Cigarettes
MeSH Terms: conditions — Tobacco Use Disorder; Smoking; Marijuana Abuse; Marijuana Smoking | interventions — Varenicline

STUDY DESIGN:
Intervention Model Description: Double Blind Placebo Controlled Trial: . Eligible individuals will be randomized to receive varenicline or matching placebo in a 1:1 manner utilizing a stratified random block design with block sizes of 2, 4 and 6.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Varenicline (Experimental): Varenicline will be provided at the standard recommended dose of 0.5mg daily for three days, then 0.5mg twice daily for four days, and then 1mg twice daily for the remainder of the 12-week treatment period.
  Interventions: Drug: Varenicline
- Placebo (Placebo Comparator): Matching placebo will be administered over the 12-week period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Varenicline — Varenicline is a selective nACHr partial agonist of the 4 2 subtype and a full agonist of the 7 subtype
  Other Names: Chantix
  Arms: Varenicline
Drug: Placebo — Matching, inactive medication
  Arms: Placebo

SUMMARY:
After initial eligibility screening, Veterans who use both cannabis and tobacco will be randomly assigned to receive either varenicline (Chantix) or placebo for 12 weeks. Participants will attend weekly visits, in person or remotely, to provide breath and urine samples for testing, fill out questionnaires, and meet with study staff about medication compliance.

DETAILED DESCRIPTION:
Screening and Eligibility Assessment. Individuals will be screened by the research study intake coordinator. An initial pre-screen focused on inclusion/exclusion psychiatric diagnoses, medical status, current medication regimen, and ability and willingness to commit to completion of study procedures will be used to initially determine potential study eligibility. Interested individuals will be given a full description of the study procedures and asked to read and sign an IRB-approved informed consent form before participating in a detailed, comprehensive screening and assessment phase.

Diagnostic/Descriptive Assessment. The MINI International Neuropsychiatric Interview (MINI) will be used to assess psychiatric and substance use diagnoses. A medical history and physical exam will be conducted to ensure that the individual is eligible to participate. In the event an individual is found to be ineligible to participate in this research protocol, he or she will be given an appropriate referral for further medical care or to an appropriate treatment program. If found eligible, a randomization visit will be scheduled, and ongoing cannabis and tobacco use will be tracked between initial assessment and randomization.

Treatment Assignment. Eligible individuals will be randomized to receive varenicline or matching placebo in a 1:1 manner utilizing a stratified random block design with block sizes of 2, 4 and 6. To achieve treatment balance, randomization will be stratified by gender and presence of comorbid psychiatric conditions (depression, PTSD, etc.) as both have been shown to modify cannabis use. The randomization allocation schedule will be developed by the study statistician (Partially blinded, A/B treatment) and all study staff, the investigative team and participants will remain blinded to study assignment until study completion or an otherwise medical necessity. The study randomization will be reviewed by the study statistician (partially blinded) on a regular basis to ensure that the schedule is being implemented according to plan. Final treatment assignment (A/B) and dispensing will be performed by the VA Investigational Pharmacy, a centralized research pharmacy that manages clinical trial medications. Varenicline will be provided at the standard recommended dose of 0.5mg daily for three days, then 0.5mg twice daily for four days, and then 1mg twice daily for the remainder of the 12-week treatment period. Medication (varenicline and matching placebo capsules) will be compounded by Pitt Street Pharmacy, a local pharmacy that has been utilized previously by VA investigators. Dr. McRae-Clark holds an IND from the FDA for the use of varenicline in individuals with cannabis use disorder.

Medication Management. Medication Management (MM) is a common-sense, generalizable approach to encourage adherence to medication specifically, and to a treatment plan in general. Once a week, participants will be seen for a brief MM session. Sessions will be focused on (a) developing and maintaining rapport, (b) reviewing AEs and concomitant medications, and (c) discussing progress with medication adherence and cannabis reduction/abstinence. These sessions provide an opportunity to address challenges and help participants devise strategies for success. In some circumstances, when patient visits are not feasible, safe, or are prohibited, such as in the case of a pandemic, MM may be completed remotely by telehealth/phone. Remote sessions will be delivered via standard desk, laptop computer, tablet, or smartphone running VA approved applications, specifically VA Video Connect/Teams.

ELIGIBILITY:
Inclusion Criteria:

* Meet DSM-5 criteria for cannabis use disorder and use cannabis at least 3 days per week in the last 30 days.
* Meet DSM-5 criteria for tobacco use disorder and smoke at least five cigarettes or report vaping 5 mg of nicotine daily.
* Males and female Veterans aged 18 and over.
* Be interested in quitting or reducing cannabis and tobacco use.
* If female and of childbearing potential, must agree to use acceptable methods of birth control for the duration of the trial.
* Must consent to random assignment, and be willing to commit to medication ingestion.
* Must be able to read and provide informed consent.
* Must have body weight >110lbs (50kg) and have BMI between 18 and 35 kg/m2
* Must function at an intellectual level and have knowledge of the English language to sufficiently allow for accurate completion of assessments.

Exclusion Criteria:

* Women who are pregnant, nursing, or plan to become pregnant during the course of the study.
* Individuals with severe renal impairment.
* Lifetime history of DSM-5 Bipolar I or II Disorder, Schizophrenia or other psychotic disorder. Stably treated MDD, Dysthymia, GAD, Social Phobia, PTSD, and Specific Phobia diagnoses are acceptable (i.e. same dose of medication/psychotherapy has been prescribed for at least 2 months prior to screening and no changes in current medication/psychotherapy expected during course of the trial).
* Suicidal ideation or behavior within the past 6 months. Subjects who are believed to be at suicidal (answers 'yes' on questions 4 or 5 of C-SSRS) or homicidal risk will be referred to assessment by a mental health professional.
* Concomitant use of psychotropic medications, with the exception of stable doses (defined as no dosing adjustments in the past two months) of non-MAO-I antidepressants, non-benzodiazepine anxiolytics, and ADHD medications.
* Current use of medications prescribed for mania or psychosis (these medications may be allowed if used for other indications)
* Current use of bupropion, amitriptyline or nortryptiline or other medication known to have drug interactions with varenicline
* Moderate or severe non-cannabis substance use disorders within the past 60 days with the exception of tobacco use disorder.
* Individuals taking an investigational agent within the last 30 days before baseline visit.
* Individuals with clinically significant medical disorders or lab abnormalities.
* Individuals with clinically significant cardiovascular disease in the past 6 months (e.g., myocardial infarction, CABG, PTCA, or severe or unstable angina).
* Individuals with clinically significant cerebrovascular disease in the past 6 months such as TIA, CVA, or stroke
* Hypersensitivity to varenicline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-04-17 (Actual); Primary Completion 2024-07-17 (Actual); Study Completion 2024-07-17 (Actual)

PRIMARY OUTCOMES:
Number of cannabis using day as reported on Timeline Followback | Weeks 6-12
  Number of cannabis using days as self-reported on TLFB
Average number cigarettes smoked per day as reported on Timeline Followback | Weeks 6-12
  Average number of cigarettes smoked per day as self-reported on TFLB

OTHER OUTCOMES:
Number of participants engaged in study visits and treatment | Week 12
  Participants will be considered retained if they are actively engaged in study visits and treatment at Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Aimee L. Mcrae-Clark, PharmD, Principal Investigator — Ralph H. Johnson VA Medical Center, Charleston, SC
Locations (1):
- Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-08-30): https://cdn.clinicaltrials.gov/large-docs/63/NCT05294263/ICF_000.pdf